CLINICAL TRIAL: NCT01304485
Title: Phase 2 Study: PET Imaging Characteristics of C11-Acetate in Patients With Prostate Carcinoma, Detection of Recurrent Disease With PSA Relapse
Brief Title: PET Imaging Characteristics of C11-Acetate in Patients With Recurrent Prostate Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Phoenix Molecular Imaging (Other)
Responsible Party: Principal Investigator, Fabio Almeida MD, Fabio Almeida MD, Medical Director, Phoenix Molecular Imaging
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AMIC-AC-001
Record Dates: First submitted 2011-02-24; First posted 2011-02-25 (Estimated); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Prostate Cancer
Keywords: Recurrent Prostate Carcinoma; sodium acetate c11; PET; prostate cancer; rising PSA; PSA recurrence; biochemical recurrence
MeSH Terms: conditions — Prostatic Neoplasms | interventions — carbon-11 acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sodium Acetate C11 PET Imaging (Experimental)
  Interventions: Drug: Sodium Acetate C11

INTERVENTIONS:
Drug: Sodium Acetate C11 — PET Imaging with Sodium Acetate C11
  Other Names: Carbon 11 Acetate PET; C11 Acetate; AC-PET

SUMMARY:
Positron emission tomography (PET) imaging evaluation in men with recurrent prostate cancer to select patients who may benefit from directed therapy

DETAILED DESCRIPTION:
The goal of this project is improved imaging of prostate cancer by positron emission tomography (PET) with use of the radiopharmaceutical C-11 Acetate, utilizing state-of-the-art PET/CT camera technology and processing algorithms.

A successful effort will lead to more accurate diagnosis of recurrence in patients with prostate cancer to allow for early directed therapy. This study is designed to generate data to add to the understanding of the effectiveness of C-11 Acetate, focusing on patients with recurrent or persistent disease after prostatectomy or radiation therapy.

The study is designed to expand on the database of C11-Acetate PET imaging in patients with prior definitive therapy for prostate cancer and evidence of biochemical recurrence (post therapy rise in PSA), and to evaluate the relationship between detection on C11-Acetate PET imaging, PSA (Trigger, Velocity and Doubling Time) and FDG PET imaging.

Specific questions to be addressed:

1. What is the yield of current state-of-the-art PET/CT with C-11 Acetate in detecting recurrent disease in this patient population?
2. How does the performance of PET with C-11 Acetate compare with that of PET using F-18 fluorodeoxyglucose (FDG-PET), Sodium F18 PET bone scans and with that of CT?
3. What is the optimal imaging protocol in terms of imaging time after injection?

ELIGIBILITY:
Inclusion Criteria:

* recurrent prostate cancer (detectable PSA following radical prostatectomy or rising PSA in patients with radiation therapy as the primary treatment)

Exclusion Criteria:

* < 18 years old
* claustrophobic patients

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Actual)
Dates: Start 2011-04; Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
SUV (Standardized Uptake Value) | Day1 - Assessed at time of PET imaging - i.e. at the time of primary investigation/PET agent administration
  Imaging studies will be evaluated both qualitatively and quantitatively using SUV (standardized uptake values): a measure of metabolism based on injected dose, patient weight and region of interest.

SECONDARY OUTCOMES:
PSA (prostate specific antigen) | Every 3 - 6 months for 24 months after PET imaging
  PSA will be monitored per routine clinical follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Almeida, M.D., Principal Investigator — Medical Director, Phoenix Molecular Imaging
Locations (1):
- Phoenix Molecular Imaging, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
Journal Publication